CLINICAL TRIAL: NCT04618146
Title: Enhanced Recovery After Cesarean Section With Low Dose Intrathecal Morphine. A Prospective Randomized Controlled Study.
Brief Title: Enhanced Recovery After Cesarean Section With Low Dose Intrathecal Morphine.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sohair Adeeb, Principle investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 680-9\2020
Record Dates: First submitted 2020-11-01; First posted 2020-11-05 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative; Pruritus; Nausea, Postoperative; Vomiting, Postoperative
Keywords: pain; morphine; cesarean section; enhanced recovery
MeSH Terms: conditions — Pain, Postoperative; Pruritus; Postoperative Nausea and Vomiting; Pain | interventions — Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): given intrathecal bupivacaine 12.5 mg.
  Interventions: Drug: Bupivacaine Hydrochloride
- Group M25 (Active Comparator): given intrathecal bupivacaine 12.5mg + morphine 25 microgram.
  Interventions: Drug: Morphine Sulfate; Drug: Bupivacaine Hydrochloride
- Group M50 (Active Comparator): given intrathecal bupivacaine 12.5mg + morphine 50 microgram.
  Interventions: Drug: Morphine Sulfate; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Morphine Sulfate — intrathecal low dose morphine for early return to normal activity without opioid related complications.
  Other Names: morphine
  Arms: Group M25; Group M50
Drug: Bupivacaine Hydrochloride — intrathecal bupivacaine 0.5%
  Other Names: marcaine

SUMMARY:
This study is designed to see the effect of low dose intrathecal morphine on promting enhanced recovery after cesarean delivery with early ambulation and reduction of hospital stay.

DETAILED DESCRIPTION:
Parturients showing for elective cesarean section will be randomized into 3 groups by a computer generated randomization list. Each randomization slip will be put in a sealed envelope until patient enrollment. Patients will be divided into Group C: control group, given intrathecal bupivacaine 12.5 mg. Group M25: intrathecal bupivacaine 12.5mg + morphine 25 microgram. Group M50: intrathecal bupivacaine 12.5mg + morphine 50 microgram.

ELIGIBILITY:
Inclusion Criteria:

* Females scheduled for cesarean section
* Age: 16-45 yrs.
* Gestation age >38 weeks.
* ASA I,II

Exclusion Criteria:

* Refusal to participate.
* Significant cardiac, hepatic or renal dysfunction.
* History of chronic itching problem, or hyperemesis during pregnancy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — females presenting for cesarean section
Enrollment: 60 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Pain postoperative | 2 hours postoperatively
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain
Pain postoperative | 4 hours postoperatively
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain
Pain postoperative | 24 hours postoperatively
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain

SECONDARY OUTCOMES:
vomiting | 2 hours postoperative
  four-point rating score (1: no nausea or vomiting, 2: queasy, 3: severe nausea, 4: vomiting).
vomiting | 4 hours postoperative
  four-point rating score (1: no nausea or vomiting, 2: queasy, 3: severe nausea, 4: vomiting).
vomiting | 24 hours postoperative
  four-point rating score (1: no nausea or vomiting, 2: queasy, 3: severe nausea, 4: vomiting).
itching | 2 hours postoperative
  four-point rating score (1: no itching, 2: mild,face, no traetment needed 3: severe itching, allover the body).
itching | 4 hours postoperative
  four-point rating score (1: no itching, 2: mild,face, no traetment needed 3: severe itching, allover the body).
itching | 24 hours postoperative
  four-point rating score (1: no itching, 2: mild,face, no traetment needed 3: severe itching, allover the body).
respiratory depression | 4 hours postoperative
  respiratory rate less than 8 breaths \ minute

CONTACTS AND LOCATIONS:
Overall Officials: Sohair A Megalla, MD, Principal Investigator — Anesthesia and ICU department, Faculty of Medicine, Minia University
Locations (1):
- Minia university, Minya, Egypt